CLINICAL TRIAL: NCT06731088
Title: Effect of Remazolam Besylate Combined With Remifentanil Analgesic Sedation on the Prognosis of Patients With Sepsis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAHNBU20241244
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam
- Remazolam benzenesulfonate (Active Comparator)
  Interventions: Drug: Remazolam besylate

INTERVENTIONS:
Drug: Midazolam — Midazolam, a benzodiazepine sedative commonly used in ICU, acts on GABA receptors in the central nervous system to produce dose-related hypnosis, anti-pyroanxiety and anterograde amnesia, and has corresponding competitive antagonists [8]. It has rapid onset and short duration, but its deficiency lies in that the metabolites are still active. Thus easy accumulation, prolong the recovery time of patients
  Arms: Midazolam
Drug: Remazolam besylate — Remazolam besylate is a new type of benzodiazepine sedative drug metabolized by tissue esterase. It is not metabolized by liver and kidney, and is metabolized by tissue esterase rapidly in vivo to produce inactive metabolites.
  Arms: Remazolam benzenesulfonate

SUMMARY:
In this study, midazolam was used as a control to investigate the effect of remazolam besylate combined with remifentanil on analgesia and sedation in patients with mechanical ventilation of sepsis on the prognosis of patients, and to provide evidence for the safe application of remazolam besylate in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical ventilation patients with sepsis who are expected to stay in ICU for ≥48h;
2. The condition was allowed to remain in shallow sedation (RASS-2 ~0);
3. Obtain informed consent from patients or family members

Exclusion Criteria:

1. pregnancy or breastfeeding;
2. General anesthesia surgery within 48 hours;
3. Severe, pre-existing parenchymatous liver disease with clinically significant portal hypertension, Child-Pugh grade C cirrhosis or acute liver failure;
4. Patients with acute and chronic renal insufficiency requiring dialysis treatment;
5. Severe craniocerebral injury, brain tumor, increased intracranial pressure, cerebrovascular accident, coma, epileptic status, etc. 6 Medical Ethics Committee of the First Affiliated Hospital of Ningbo University;
6. Patients with a history of alcohol or drug abuse;
7. Any condition that prevents the correct assessment of cognitive function, such as speech and sensory disorders or mental disorders (language difficulties or organic mental dysfunction);
8. Failure to obtain informed consent or authorization;
9. Participate in other exploratory clinical trials within 6 months prior to screening;
10. Known or suspected allergy to the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of days without delirium or coma during the 14-day intervention period. | From enrollment to the end of treatment at 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China